CLINICAL TRIAL: NCT03956836
Title: Perioperative Coagulopathy in Patients Undergoing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Brief Title: Perioperative Coagulopathy in Patients Undergoing Cytoreductive Surgery and HIPEC Intraperitoneal Chemotherapy (HIPEC)
Acronym: HIPEC-COAG
Status: Completed | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Antonio M. Puppo Moreno, Critical Care Staff, Hospitales Universitarios Virgen del Rocío
Other Study IDs: HUVirgenRocio
Record Dates: First submitted 2019-05-13; First posted 2019-05-21 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Coagulation Disorder; Carcinomatosis
MeSH Terms: conditions — Hemostatic Disorders; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ROTEM parameters, platelet function assay (PFA-100), von Willebrand and Factor XIII — ROTEM parameters, platelet function assay (PFA-100), von Willebrand and Factor XIII at baseline (before surgery) and after 4h and 48 after surgery in 40 patients undergoing CRC
  Other Names: ROTEM, PFA-100

SUMMARY:
Cytoreductive surgery (CRC) with intraperitoneal hyperthermal chemotherapy (HIPEC) has been shown to improve survival in selected patients with peritoneal carcinomatosis. 51% of patients are transfused due to the high intraoperative blood loss caused by surgery and the appearance of a perioperative coagulopathy attributed to the loss of proteins into the peritoneal cavity, the high fluid turnover and possibly the action of hyperthermic chemotherapy. So far, the haemostatic changes described consist of a decrease in the levels of antithrombin III and the platelet count, as well as in alterations of the usual coagulation tests. Conventional coagulation tests analyze only the plasmatic phase of coagulation while viscoelastic tests, such as rotational thromboelastometry (ROTEM), reproduce the global coagulation process much more faithfully, keeping good correlation with perioperative bleeding.

Objetive:

The platelet, coagulation, von Willebrand and Factor XIII levels and function have not been consistently investigate in pre-established (fix) time periods in patients undergoing elective CRC with hyperthermia. This prospective observational study aimed at investigating the variations of the values of estándar coagulation test, ROTEM parameters, platelet function assay (PFA-100), von Willebrand and Factor XIII at baseline (before surgery) and after 4h and 48 after surgery in 40 patients undergoing CRC. A control group (N=40 blood donors) will be also obtained by baseline comparasion and to obtain local reference ranges.

DETAILED DESCRIPTION:
This prospective observational study aimed at investigating the variations of the values of estándar coagulation test, ROTEM parameters, platelet function assay (PFA-100), von Willebrand and Factor XIII at baseline (before surgery) and after 4h and 48 after surgery in 40 patients undergoing CRC. A control group (N=40 blood donors) will be also obtained by baseline comparasion and to obtain local reference ranges.

ELIGIBILITY:
Inclusion Criteria:

1. - Consecutive patients with peritoneal surface malignancy treated with cytoreductive surgery and HIPEC in the Department of Surgery of Virgen del Rocio General Hospital
2. -All patients gave written informed consent.
3. -Age above 18 years and Karnofsky performance status scale 450%

Exclusion Criteria:

1. - Exclusion criteria: were severe cardiovascular or respiratory disease,
2. - Lower hemoglobin than 10,0 g/dL , platelet count 100,000/mm3,
3. - Renal or hepatic failure,
4. - Pregnancy,
5. - Multiple partial intestinal obstruction or extensive involvement of the surface of the small bowel as well as distant and non-resectable metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of peritoneal surface malignancy of the ovarian and/or colo origin undergoing complete cytoreductive surgery (zero) combined with Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Variations of CT-ROTEM | 48 hours
  variations in clotting time of ROTEM from baseline (preoperative) to 48 hours post surgery
Variations of MCF-ROTEM | 48 hours
  variations in maximum clotting firmness of ROTEM 48 hours post surgery
Variations of PFA-100 | 48 hours
  variations in COL-EPI (platelet function) from of 48 hours post surgery
Variations of Factor XIII | 48 hours
  variations in factor XIII Concentration of clotting factor from baseline (preoperative) of 48 hours post surgery
Variations of von Willebrand | 48 hours
  variations in von Willebrand Concentration from 48 hours post surgery

SECONDARY OUTCOMES:
Transfusion of red blood cells | 20 days
  number of packed red blood cells and percentage of transfused patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No